CLINICAL TRIAL: NCT00192712
Title: Phase II Study of Irinotecan and Gemcitabine (IrinoGem) Combined With 3-D Conformal Radiation Therapy for Locally Advanced Pancreatic Cancer
Brief Title: Irinotecan, Gemcitabine and Radiation Therapy for Pancreatic Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RonIrinoGem.CTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-09

CONDITIONS: Pancreatic Cancer
Keywords: carcinoma; pancreas; chemotherapy; radiotherapy
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma | interventions — Irinotecan; Gemcitabine

INTERVENTIONS:
Drug: irinotecan, gemcitabine

SUMMARY:
The study hypothesis is that chemoradiation based on 2 drugs will improve local control and long-term survival in patients with locally advanced pancreatic cancer. That is why gemcitabine and irinotecan are combined in an induction phase of 2 months and then this IrinoGem combination is given for 3 more cycles, in reduced doses,concurently with irradiation.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced pancreatic cancer
* performance status 0-2
* normal blood count and chemistry
* no previous chemotherapy or radiotherapy

Exclusion Criteria:

* serious concurrent systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-11; Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
time to treatment failure

SECONDARY OUTCOMES:
response rate, survival, toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ron Epelbaum, MD, Principal Investigator
Locations (1):
- Department of Oncology, Rambam Medical Center, Haifa, Israel